CLINICAL TRIAL: NCT00627679
Title: A Randomized, Double Blind, Active Controlled, Single Dose, 4 Arm, 4 Period Crossover, Phase 1 Study Investigating the Tolerability and Pharmacokinetics of MAP0010
Brief Title: Safety and Blood Level Study of Unit Dose Budesonide
Acronym: UDB P101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry); Q-Pharm Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MAP0010-CL-P101
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: Pediatric asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment sequence: A, B, D, C (Experimental): Treatment visits were separated by a 48-72 hour washout period. Treatment A = a single dose of Budesonide inhalation suspension (Pulmicort Respules®) delivered by nebulization at Visit 2; Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 3; Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 4; Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 5
  Interventions: Drug: Budesonide Inhalation Suspension; Drug: MAP0010 low dose; Drug: MAP0010 intermediate dose; Drug: MAP0010 high dose
- Treatment sequence: B, C, A, D (Experimental): Treatment visits were separated by a 48-72 hour washout period. Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 2; Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 3; Treatment A = a single dose of Budesonide inhalation suspension (Pulmicort Respules®) delivered by nebulization at Visit 4; Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 5
  Interventions: Drug: Budesonide Inhalation Suspension; Drug: MAP0010 low dose; Drug: MAP0010 intermediate dose; Drug: MAP0010 high dose
- Treatment sequence: C, D, B, A (Experimental): Treatment visits were separated by a 48-72 hour washout period. Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 2; Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 3; Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 4; Treatment A = a single dose of Budesonide inhalation suspension (Pulmicort Respules®) delivered by nebulization at Visit 5
  Interventions: Drug: Budesonide Inhalation Suspension; Drug: MAP0010 low dose; Drug: MAP0010 intermediate dose; Drug: MAP0010 high dose
- Treatment sequence: D, A, C, B (Experimental): Treatment visits were separated by a 48-72 hour washout period. Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 2; Treatment A = a single dose of Budesonide inhalation suspension (Pulmicort Respules®) delivered by nebulization at Visit 3; Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 4; Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 5
  Interventions: Drug: Budesonide Inhalation Suspension; Drug: MAP0010 low dose; Drug: MAP0010 intermediate dose; Drug: MAP0010 high dose

INTERVENTIONS:
Drug: Budesonide Inhalation Suspension — Treatment A = a single dose of Pulmicort Respules® (budesonide inhalation suspension) delivered by nebulization at Visit 2, 3, 4, or 5 as per protocol.
  Other Names: Pulmicort Respules®
Drug: MAP0010 low dose — Treatment B = a single dose of MAP0010 (unit dose budesonide) low dose delivered by nebulization at Visit 2, 3, 4, or 5 as per protocol.
Drug: MAP0010 intermediate dose — Treatment C = a single dose of MAP0010 (unit dose budesonide) intermediate dose delivered by nebulization at Visit 2, 3, 4, or 5 as per protocol.
Drug: MAP0010 high dose — Treatment D = a single dose of MAP0010 (unit dose budesonide) high dose delivered by nebulization at Visit 2, 3, 4, or 5 as per protocol.

SUMMARY:
The purpose of this study is to evaluate the tolerability and pharmacokinetics of three doses of MAP0010 (Unit Dose Budesonide) compared with Pulmicort Respules® (Budesonide) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, aged 18-50 years
* BMI less than 30 kg/m2
* Non smoker (currently and <10 pack years total if ex-smoker)

Exclusion Criteria:

* Any use of corticosteroid in previous 4 weeks
* Pregnancy/lactation
* Significant blood donation (or testing) in previous 8 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-12; Primary Completion 2005-12 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Marjason, MBBS, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Q-Pharm Pty Limited, Brisbane, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects received all 4 treatments in a randomly assigned order. The treatments were:
  Treatment A: Pulmicort Respules® Treatment B: MAP0010 low dose Treatment C: MAP0010 intermediate dose Treatment D: MAP0010 high dose The sequences were Treatments ABDC, BACD, CDBA, DACB.
Groups:
- Treatment A, B, D, C: Treatment visits were separated by a 48-72 hour washout period. Treatment A = a single dose of Pulmicort Respules® delivered by nebulization at Visit 2; Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 3; Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 4; Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 5
- Treatment B, C, A, D: Treatment visits were separated by a 48-72 hour washout period. Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 2; Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 3; Treatment A = a single dose of Pulmicort Respules® delivered by nebulization at Visit 4; Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 5
- Treatment C, D, B, A: Treatment visits were separated by a 48-72 hour washout period. Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 2; Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 3; Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 4; Treatment A = a single dose of Pulmicort Respules® delivered by nebulization at Visit 5
- Treatment D, A, C, B: Treatment visits were separated by a 48-72 hour washout period. Treatment D = a single dose of MAP0010 high dose delivered by nebulization at Visit 2; Treatment A = a single dose of Pulmicort Respules® delivered by nebulization at Visit 3; Treatment C = a single dose of MAP0010 intermediate dose delivered by nebulization at Visit 4; Treatment B = a single dose of MAP0010 low dose delivered by nebulization at Visit 5
Period: Overall Study
Arm/Group | Treatment A, B, D, C | Treatment B, C, A, D | Treatment C, D, B, A | Treatment D, A, C, B
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients that were enrolled in the study.
Arm/Group | All Patients
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Cmax of of Budesonide After Administration of Pulmicort and Three Dose Levels of MAP0010
Description: The maximum concentration (Cmax) is the highest concentration of a drug measured in the plasma. Plasma is the clear portion of the blood. The Cmax of Budesonide is reported in picograms per milliliter (pg/ml).
Time Frame: 8 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Treatment A: a single dose of Pulmicort Respules® delivered by nebulization as per protocol
- Treatment B: a single dose of MAP0010 low dose delivered by nebulization as per protocol
- Treatment C: a single dose of MAP0010 intermediate dose delivered by nebulization as per protocol
- Treatment D: a single dose of MAP0010 high dose delivered by nebulization as per protocol
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 15 | 16 | 16
pg/mL | 303.5 (177.4) | 106.2 (63.47) | 239.9 (140.1) | 434.5 (246.9)

2. Primary Outcome: Tmax of Budesonide After Administration of Pulmicort Respules® and Three Dose Levels of MAP0010
Description: Tmax is the time to maximum concentration of a drug in the plasma. The Tmax of budesonide is reported in minutes (min).
Time Frame: 8 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 15 | 16 | 16
min | 9.063 (7.122) | 4.467 (3.270) | 3.125 (1.500) | 3.688 (1.448)

3. Primary Outcome: AUC(0-8) of Budesonide After Administration of Pulmicort Respules® and Three Doses of MAP0010
Description: The AUC(0-8) is the area under the plot of plasma concentration of drug against time after drug administration. Budesonide AUC(0-8) is reported in picograms times minutes per milliliter (pg*min/ml).
Time Frame: 8 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 15 | 16 | 16
pg*min/mL | 29040 (9316) | 3978 (1974) | 8626 (4184) | 22130 (9675)

4. Primary Outcome: AUC(0-inf) of Budesonide After Administration of Pulmicort Respules® and Three Dose Levels of MAP0010
Description: The AUC(0-inf) is the area under the plot of plasma concentration of drug against time to infinity (inf) after drug administration. Budesonide AUC(0-inf) is reported in picograms times minutes per milliliter (pg*min/ml).
Time Frame: 8 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 12 | 13 | 14
pg*min/mL | 31480 (10690) | 4391 (1423) | 7842 (3647) | 25290 (11750)

5. Primary Outcome: Half-life (t1/2) of Budesonide After Administration of Pulmicort Respules® and Three Dose Levels of MAP0010
Description: Half-life (t1/2) is the time for the drug to decrease to half of its maximum concentration. Budesonide t1/2 is reported in minutes (min).
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 12 | 13 | 14
min | 145.4 (40.84) | 73.02 (33.43) | 78.35 (27.08) | 140.0 (54.19)

ADVERSE EVENTS:
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 4/16 | 3/16 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=16) | Treatment B (N=16) | Treatment C (N=16) | Treatment D (N=16)
thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
hematoma (Vascular disorders) | 0 | 0 | 0 | 1
epitaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
headache (Nervous system disorders) | 0 | 1 | 0 | 0
herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
vaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
anemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
eye irritation (Eye disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.